CLINICAL TRIAL: NCT00166088
Title: Effects of Mediterranean Diet and Omega-3 Fatty Acids on Oxidative Stress and EPC's
Brief Title: Effect of a Mediterranean Diet and Omega-3 Fatty Acids on Oxidative Stress and Endothelial Progenitor Cells (EPC's)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0020-2005
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Obesity
Keywords: Oxidative Stress; Diet, Mediterranean
MeSH Terms: conditions — Obesity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mediterranean Diet Arm (Experimental)
  Interventions: Dietary Supplement: Mediterranean Diet
- Mediterranean Dietary Supplement Arm (Active Comparator)
  Interventions: Dietary Supplement: Mediterranean Dietary Supplement
- Control Arm (No Intervention)

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet — The Mediterranean diet group will receive all meals as a prototypical Mediterranean diet for 4 consecutive weeks prepared by the GCRC metabolic kitchen with dietary instruction. During the second month of the study they will be asked to follow a Mediterranean diet using their own home-cooked meals
  Arms: Mediterranean Diet Arm
Dietary Supplement: Mediterranean Dietary Supplement — The subjects randomized to the typical diet + targeted Mediterranean dietary supplement group will not receive dietary counseling. They will be given a one-month supply of specific supplements by the GCRC nutritionists and advised to consume these daily, in addition to their usual diet.
  Arms: Mediterranean Dietary Supplement Arm

SUMMARY:
Problem of Interest:

A typical American diet that is high in an intake of fats (especially saturated fats and cholesterol) is known to lead to high blood levels of cholesterol, hardening of the arteries, and increases the risk of heart disease. The American Heart Association recommendations to follow a diet that is low in the amount of fat, and specifically cholesterol, that is eaten can improve blood levels of cholesterol but can lead to a high intake of sugars (especially processed sugars) that can lead to obesity and continued heart problems.

Studies of people who eat a diet that is typical of the Mediterranean region have shown that this type of diet leads to reductions in heart disease as well as forms of cancer. A typical Mediterranean diet has a large amount of fruit, vegetables, whole grain breads and cereals, beans, potatoes and seeds. Olive oil is the main source of fat and there is a daily use of dairy products (such as cheese and yogurt) in low to moderate amounts. The main meats are fish or poultry with rare red meat. Desserts are usually fruits with rare sweets. Wine is also used in low to moderate amounts with meals.

No isolated aspect of the diet explains all of its benefits, but it is believed that the ingredient of the diet that most helps to reduce the risk of heart disease is the high amount of omega-3 fatty acids. Omega-3 fatty acids are found in fatty fish as well as in nuts and certain oils. Several studies of patients with either known heart disease or risk factors for heart disease have shown a reduction in heart disease events, such as heart attacks, as well as markers of heart disease risk when patients followed a Mediterranean diet. Other studies have shown that giving a supplement that contains omega-3 fatty acids to patients with heart disease or risk factors for heart disease also reduces heart disease events and markers of heart disease risk.

In this current study we, the investigators at Emory University, plan to compare the effects of following a Mediterranean diet versus continuing to follow an American type diet and supplementing parts of the Mediterranean diet, including omega-3 fatty acids, on markers of heart disease risk. A third group will continue to follow their usual diet without supplements to serve as a control.

How Problem Will be Studied:

In this initial study we will compare three groups. One group will receive one month of prepared meals that will follow a Mediterranean diet. This group will also receive extensive counseling and education on how to maintain a Mediterranean diet. During the second month of the study this group will be encouraged to continue following a Mediterranean diet by themselves with assistance from a nutritionist. The second group will be asked to continue on their current diet and receive supplements that are important parts of the Mediterranean diet. These supplements will include an omega-3 fatty acid capsule, walnuts and grape juice. A third group will be asked to continue their current diet and level of activity without supplements to serve as a control. We will follow the effects on markers of heart disease risk. We will also determine if patients are able to continue following a Mediterranean diet on their own or whether simply taking supplements is easier.

Advancement in Scientific Knowledge:

This study will advance scientific knowledge by comparing the effects of following a Mediterranean diet versus simply taking supplements of the believed to be important aspects of the Mediterranean diet. We will also be able to determine if it is easier to follow a Mediterranean diet or take supplements for patients who are currently ingesting a typical American diet.

Standard of Care:

Currently the recommended diet for all Americans is a Step 1 American Heart Association diet that is low in fat and specifically low in saturated fats and cholesterol. As stated above, despite these recommendations, there is a growing problem of obesity in the United States and there is evidence to suggest that a Mediterranean diet may be better.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [BMI; body weight (kg)/height (m)2] greater than or equal to 28 and less than 35
* Stable body weight in the past 6 months (weight change < 2 kg)
* Non-smokers
* Currently consuming a stable habitual diet as assessed by interview with a nutritionist and 24 hour diet recall showing:

  * saturated + trans fat intake of > 10% of total daily calories; and
  * total cholesterol intake of > 300 mg/day
* Not consuming antioxidants or vitamin-mineral preparations in the last 4 weeks

Exclusion Criteria:

* History of significant cardiovascular disease
* Cancer other than remote history of skin cancer
* Diabetes mellitus by history or fasting plasma glucose (FPG) > 126mg/dL
* Excessive chronic alcohol consumption (averaging > two alcoholic beverages/day)
* Known acute or chronic illness, including psychiatric problems that will, in the opinion of the principal investigator (PI), make one ineligible for the study
* Statin or other hypolipidemic therapy
* Current intake of vitamins and supplements
* Inability to return to Emory for follow-up, blood drawing
* Pregnant or lactating females
* Unable to give informed consent
* Hematocrit < 30%
* Uncontrolled hypertension with systolic blood pressure (SBP) > 180 and diastolic blood pressure (DBP) > 110
* History of bleeding disorder

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Brachial artery reactivity to test flow-mediated vasodilation (FMD) as a measure of endothelial function. | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States